CLINICAL TRIAL: NCT00155987
Title: Multi-centre Prospective Randomised Trial of Early Decompressive Craniectomy in Patients With Severe Traumatic Brain Injury
Brief Title: The DECRA Trial: Early Decompressive Craniectomy in Patients With Severe Traumatic Brain Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Trauma Research Institute (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Victorian Trauma Foundation (Other); ANZICS Foundation (Other); Western Australian Institute for Medical Research (Other)
Responsible Party: Principal Investigator, Prof Jamie Cooper, Chief Investigator, National Trauma Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 68/02
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Brain Injuries
Keywords: Severe diffuse TBI refractory intracranial hypertension.
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Early decompressive craniectomy — Large bifrontotemporal decompressive craniectomy

SUMMARY:
This is a multi-centre randomised trial to evaluate the effect of early decompressive craniectomy on neurological function in patients with severe traumatic brain injury.

The primary outcome is neurological function measured at 6 months post injury using the Glasgow Outcome Score. Neurological function is qualified as proportion of favourable outcomes (Glasgow Outcome Score Extended [GOSE] grades 5-8).

DETAILED DESCRIPTION:
Comparison After meeting the entry criteria, and the patient will be randomised to either early DC surgery (see below) or best current conventional management. Those randomised to surgery will have the operation done within 6 hours of randomisation. They will then return to the ICU and be managed thereafter in the same way as the conventional arm. Patients in the conventional arm will have all the usual therapies for increasing ICP optimised again. They then may have cooling to 35.0C or thiopentone bolus or thiopentone coma. These options are at the clinicians discretion. Late DC surgery in the control patients is discouraged however it may be done at the neurosurgeons discretion. These patients will be included in the intention to treat analysis.

Surgical Technique The technique described by Polin will be used. The operation will comprise bi-frontal decompressive craniectomies with a single fronto-temporal bone flap extending across the midline. The temporalis muscles will be reflected inferiorly. Burr holes are located either side of the sagittal sinus at the posterior extent and bilaterally at the keyhole and at the root of the zygoma. This will create a large bifrontal craniectomy defect extending posteriorly to the coronal sutures. Bilateral large sub-temporal decompressions will be performed down to the skull base. The final bone cut is made along the supra-orbital ridges with an attempt to preserve the frontal sinus. Burr holes will be placed either side of the sagittal sinus inferiorly and the bone will be lifted out.

The dura will be opened in one of two alternative ways:

1. The dura is opened with a cruciate incision bilaterally. OR
2. A large L shaped incision with the lower corner of the L facing laterally. The advantage to this method is that the cerebral veins are not disturbed medially by this incision.

The dural opening should be covered with a dural or facial patch, so that the brain does not adhere to the scalp. Water tight dural closure is not necessarily aimed for. For patients receiving EVD monitoring, an ICP monitor with ventricular catheter (± optional PO2 and temperature monitor) may be placed prior to closure. Some patients will have been randomised to parenchymal catheter only. These patients will not have an EVD inserted.

The bone flap is replaced once bone swelling has resolved and the patient has improved and left the intensive care unit (6-12 weeks). The bone flap is stored at minus 20o-70oC until reinsertion or it may be implanted in the subcutaneous tissue of the abdominal wall as an alternative.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 - 60 years and within the first 72 hrs from time of injury
* Severe diffuse Traumatic Brain Injury defined as:
* GCS < 9 and CT scan* with any evidence of brain swelling CT brain scan (DII + some evidence of swelling or DIII or DIV) OR
* GCS >8 before intubation and DIII or DIV CT brain scan (basal cistern compression ± midline shift)
* ICP monitor in situ. EVD recommended.
* "Refractory ICP" despite best conventional management. Refractory ICP in this study will be defined as the spontaneous persistent increase in ICP despite optimal conventional ICU therapies (including intermittent EVD venting) of >20mm Hg for more than 15 mins (continuously or cumulative over one hour).

Exclusion criteria:

* Intracranial haemorrhage > 3 cm diameter
* Intracranial mixed haemorrhagic contusion >5cm in long axis
* Previous craniectomy
* EDH/SDH/ or large contusion requiring evacuation
* EDH/SDH >0.5 cm thickness
* Spinal cord injury
* Penetrating brain injury
* Arrest at scene
* Unreactive pupils >4mm, and GCS=3
* Neurosurgery contraindicated (eg: severe coagulopathy)
* No chance of survival after consideration of CT and clinical findings following Neurosurgical consultant assessment (eg hemispheric infarct after carotid dissection).

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 155 (Actual)
Dates: Start 2003-08; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Proportion (%) of favourable outcomes (GOSE 5-8) | 6 month post injury

SECONDARY OUTCOMES:
Mean and maximum hourly intracranial pressure (ICP) | 36hrs post randomisation
Favourable outcomes (GOSE) | 12 months post injury
Mean GOSE using ordinal logistic regression | 6 months and 12 months
Mortality | hospital, 6 months, 12 months
length of stay | ICU admisssion
Brain metabolites using microdialysis (The Alfred Hospital only) | During monitoring phase

CONTACTS AND LOCATIONS:
Overall Officials: D. J. Cooper, Principal Investigator — The Alfred Hospital & National Trauma Research Institute
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia